CLINICAL TRIAL: NCT04524364
Title: Pulsed Field Ablation (PFA) System for the Treatment of Paroxysmal Atrial Fibrillation (PAF) by Irreversible Electroporation (IRE)
Brief Title: A Study for Treatment of Paroxysmal Atrial Fibrillation (PAF) by Pulsed Field Ablation (PFA) System With Irreversible Electroporation (IRE)
Acronym: inspIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI_2019_08; BWI_2019_08 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Participants with Paroxysmal Atrial Fibrillation (PAF) (Other): Participants with PAF and who are candidates for catheter ablation will be enrolled.
  Interventions: Device: Pulsed Field Ablation (PFA) Therapy

INTERVENTIONS:
Device: Pulsed Field Ablation (PFA) Therapy — Participants will undergo PFA therapy with a compatible ablation catheter when used with Multi-Channel irreversible electroporation (IRE) Generator (deliver trains of high-voltage bipolar pulses of short duration on separate channels to a multi-electrode ablation catheter) and Circular IRE Catheter (indicated for use in catheter-based cardiac electrophysiological mapping (stimulating and recording) and, when used with an IRE Generator, for cardiac ablation).

SUMMARY:
The primary objective is to demonstrate safety and long-term effectiveness of the irreversible electroporation (IRE) system (Circular IRE Catheter and IRE Generator) when used for isolation of the atrial pulmonary veins (PVs) in treatment of participants with paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Symptomatic paroxysmal atrial fibrillation (PAF)
* Selected for atrial fibrillation (AF) ablation procedure by pulmonary vein isolation (PVI)
* Failed at least one antiarrhythmic drug (AAD) (class I to IV) as evidenced by recurrent symptomatic atrial fibrillation AF, or intolerable or contraindicated to the AAD
* Willing and capable of providing consent
* Able and willing to comply with all pre-, post- and follow-up testing and requirements

Exclusion Criteria:

* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Previous left atrium (LA) ablation or surgery
* Participant known to require ablation outside the PV region (example. cavotricuspid isthmus [CTI] region, atrioventricular reentrant tachycardia, atrioventricular nodal reentry tachycardia, atrial tachycardia, ventricular tachycardia and Wolff-Parkinson-White)
* Previously diagnosed with persistent AF (greater than [>] 7 days in duration)
* Severe dilatation of the LA (LAD >50 millimeter (mm) antero-posterior diameter in case of transthoracic echocardiography (TTE))

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2020-08-23 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Austria (2):
  - Medical University Graz, Graz
  - Ordensklinikum Linz Elisabethinen, Linz
- Belgium (4):
  - OLV Aalst, Aalst
  - AZ Sint-Jan Brugge, Bruges
  - Ziekenhuis Oost-Limburg Genk Campus Sint-Jan, Genk
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket
- University Hospital Center Split, Split, Croatia
- Nemocnice na Homolce, Prague, Czechia
- Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux, France
- Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti, Italy
- Vilnius University Hospital, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.

REFERENCES:
- [Derived] De Potter T, Grimaldi M, Duytschaever M, Anic A, Vijgen J, Neuzil P, Van Herendael H, Verma A, Skanes A, Scherr D, Purerfellner H, Rackauskas G, Jais P, Reddy VY; inspIRE Trial Investigators. Predictors of Success for Pulmonary Vein Isolation With Pulsed-field Ablation Using a Variable-loop Catheter With 3D Mapping Integration: Complete 12-month Outcomes From inspIRE. Circ Arrhythm Electrophysiol. 2024 May;17(5):e012667. doi: 10.1161/CIRCEP.123.012667. Epub 2024 Apr 24. PMID 38655693
- [Derived] Duytschaever M, De Potter T, Grimaldi M, Anic A, Vijgen J, Neuzil P, Van Herendael H, Verma A, Skanes A, Scherr D, Purerfellner H, Rackauskas G, Jais P, Reddy VY; inspIRE Trial Investigators. Paroxysmal Atrial Fibrillation Ablation Using a Novel Variable-Loop Biphasic Pulsed Field Ablation Catheter Integrated With a 3-Dimensional Mapping System: 1-Year Outcomes of the Multicenter inspIRE Study. Circ Arrhythm Electrophysiol. 2023 Mar;16(3):e011780. doi: 10.1161/CIRCEP.122.011780. Epub 2023 Feb 3. PMID 36735937

RESULTS

PARTICIPANT FLOW:
Groups:
- Wave I: Participants with drug refractory, symptomatic pulse field ablation (PAF) who were candidates for catheter ablation, underwent the index procedure and additional neurological, pulmonary vein (PV) and esophageal assessments to obtain data for preliminary estimates of safety and (acute) effectiveness of the irreversible electroporation (IRE) ablation system.
- Wave II: Participants were enrolled in Wave II (Wave II main phase or Wave II roll-in) and treated with the Circular IRE Catheter in conjunction with the IRE Generator.
Period: Overall Study
Arm/Group | Wave I | Wave II
Started | 45 | 227
Treated | 40 | 216
Wave II: Main Phase Full Analysis Set | 0 | 186
Wave II: Roll-in Analysis Set (RI AS) | 0 | 30
Completed | 40 | 216
Not Completed | 5 | 11
Not completed — Physician Decision | 3 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Investigational device deficiency | 0 | 1
Not completed — Implantable cardioverter device (ICD) discovered | 0 | 1
Not completed — Device unavailability | 0 | 2
Not completed — Atrio-ventricular Paroxysmal tachycardia requiring ablation outside PV | 1 | 0
Not completed — Low International normalized ratio (INR) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were based on the full analysis set (FAS) for Wave I and Wave II (main phase) arms and the roll-in analysis set (RI AS) for the Wave II (roll-in) arm. FAS included all enrolled Wave I and Wave II (main phase) participants who had insertion of the study catheter (with or without delivery of PFA). The RI AS included all Wave II (roll-in) participants who were enrolled in the roll-in phase and underwent ablation with the irreversible electroporation (IRE) ablation system.
Groups:
- Wave II: Main Phase: Participants enrolled in Wave II main phase, were treated with the Circular IRE Catheter in conjunction with the IRE Generator.
- Wave II: Roll-In: Participants enrolled in Wave II roll-in, were treated with the Circular IRE Catheter in conjunction with the IRE Generator.
- Total: Total of all reporting groups
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In | Total
Number analyzed (Participants) | 40 | 186 | 30 | 256
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (10.86) | 59.4 (10.18) | 56.2 (11.72) | 58.0 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 55 | 10 | 82
  Male | 23 | 131 | 20 | 174
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Adverse Events (PAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. The primary safety endpoint was the incidence of PAEs (within 7 days of the initial mapping and ablation procedure). PAEs included the following AEs: Atrio-esophageal fistula, cardiac tamponade/perforation, device or procedure related death, major vascular access complication/bleeding, myocardial infarction, pericarditis, phrenic nerve paralysis (permanent), pulmonary vein stenosis, stroke/cerebrovascular accident (CVA), thromboembolism, and transient ischemic attack (TIA).
Time Frame: Within 7 days post-procedure on Day 0
Population: Wave I and Wave II (Main Phase): The full analysis set (FAS) included all enrolled Wave I and Wave II (main phase) participants who had insertion of the study catheter (with or without delivery of pulse field ablation [PFA]); Wave II (Roll-in): The Roll-In analysis set (RI AS) included all Wave II (roll-in) participants who were enrolled in the roll-in phase and underwent ablation with the irreversible electroporation (IRE) ablation system.
Measure: Count of Participants; unit: Participants
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In
Number analyzed (Participants) | 40 | 186 | 30
Participants | 0 | 0 | 0

2. Primary Outcome: Kaplan-Meier Estimates of the Success Rate of Freedom From Documented (Symptomatic and Asymptomatic) Atrial Arrhythmia (Atrial Fibrillation [AF], Atrial Tachycardia [AT], or Atrial Flutter [AFL]) Episodes From Day 91 to Day 365 Post Index Procedure
Description: Kaplan-Meier estimates of the success rate of freedom from primary effectiveness failure, that is, documented (symptomatic and asymptomatic) atrial arrhythmia (AF, AT, or AFL) recurrence based on electrocardiographic data (>=30 seconds on arrhythmia monitoring device) from Day 91 to Day 365 post index procedure, was reported. Acute procedural failure defined as failure to confirm entrance block in all PVs except those that are silent and/or cannot be cannulated post-procedure, use of a non-study catheter for PV isolation, or failure to have PFA delivery with the study catheter due to IRE system malfunctions, was also considered a long-term effectiveness failure.
Time Frame: From Day 91 up to Day 365 post index procedure on Day 0
Population: Wave I and Wave II (Main Phase): The FAS included all enrolled Wave I and Wave II (main phase) participants who had insertion of the study catheter (with or without delivery of PFA); Wave II (Roll-in): The RI AS included all Wave II (roll-in) participants who were enrolled in the roll-in phase and underwent ablation with the IRE ablation system.
Measure: Number; unit: Percentage of participants
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In
Number analyzed (Participants) | 40 | 186 | 30
Percentage of participants | 71.8 | 75.6 | 80.0

3. Secondary Outcome: Number of Participants Who Achieved Acute Procedural Success
Description: Number of participants who achieved acute procedural success were reported. Acute procedural success was defined as confirmation of entrance block in all clinically relevant targeted pulmonary veins (PVs) after adenosine/ isoproterenol challenge.
Time Frame: Day 0 (Day of procedure)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In
Number analyzed (Participants) | 40 | 186 | 30
Participants | 40 | 186 | 30

4. Secondary Outcome: Kaplan-Meier Estimates of the Success Rate of Freedom From Documented Symptomatic Re-Occurrence of Atrial Arrhythmia (Atrial Fibrillation [AF], Atrial Tachycardia [AT], or Atrial Flutter [AFL]) Episodes From Day 91 to Day 365 Post Index Procedure
Description: Kaplan-Meier estimates of the success rate of freedom from primary effectiveness failure, that is, documented symptomatic re-occurrence of atrial arrhythmia (AF, AT, or AFL) episodes based on electrocardiographic data (>=30 seconds on arrhythmia monitoring device) from Day 91 to Day 365 post index procedure, was reported. Acute procedural failure defined as failure to confirm entrance block in all PVs except those that are silent and/or cannot be cannulated post-procedure, use of a non-study catheter for PV isolation, or failure to have PFA delivery with the study catheter due to IRE system malfunctions, was also considered a long-term effectiveness failure.
Time Frame: From Day 91 up to Day 365 post index procedure on Day 0
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In
Number analyzed (Participants) | 40 | 186 | 30
Percentage of participants | 76.9 | 81.7 | 80.0

5. Secondary Outcome: Change From Baseline in Atrial Fibrillation Effect on Quality of Life (AFEQT) Total Score
Description: Change from baseline in AFEQT total score was reported. The AFEQT questionnaire is an atrial fibrillation-specific health-related quality of life (HRQoL) questionnaire designed to assess the impact of atrial fibrillation on participants' HRQoL. The questionnaire includes 20 questions on a 7-point Likert scale. Questions 1-18 evaluate HRQoL and questions 19-20 relate to participants' satisfaction with treatment. Overall or subscale scores range from 0 to 100, where 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered). Therefore, a positive change in score corresponds to improvement in QoL. Total score was calculated using AFEQT formula: 100 -([sum of severity for all questions answered - number of questions answered]*100 / total number questions answered*6).
Time Frame: Baseline, Months 3, 6, and 12
Population: The FAS included all enrolled Wave I and Wave II (main phase) participants who had insertion of the study catheter (with or without delivery of PFA). The RI AS included all Wave II (roll-in) participants who were enrolled in the roll-in phase and underwent ablation with the IRE ablation system. Here, 'N' (number of participants analyzed) indicates number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed for specified timepoints.
Measure: Mean (Standard Deviation); unit: Units on a score
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In
Number analyzed (Participants) | 35 | 182 | 24
Units on a score
  Month 3 | 27.38 (19.685) | 23.02 (22.755) | 26.03 (22.693)
  Month 6: number analyzed (Participants) | 34 | 182 | 24
  Month 6 | 28.21 (16.422) | 25.06 (20.793) | 24.77 (23.414)
  Month 12: number analyzed (Participants) | 35 | 176 | 24
  Month 12 | 30.5 (19.897) | 26.05 (21.642) | 31.17 (19.723)

ADVERSE EVENTS:
Time Frame: From screening up to 12 months
Description: Wave I and Wave II (Main Phase): The full analysis set (FAS) included all enrolled Wave I and Wave II (main phase) participants who had insertion of the study catheter (with or without delivery of pulse field ablation [PFA]); Wave II (Roll-in): The Roll-In analysis set (RI AS) included all Wave II (roll-in) participants who were enrolled in the roll-in phase and underwent ablation with the irreversible electroporation (IRE) ablation system.
Arm/Group | Wave I | Wave II: Main Phase | Wave II: Roll-In
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/186 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/40 | 9/186 | 2/30
Other Adverse Events (participants affected / at risk) | 30/40 | 85/186 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wave I (N=40) | Wave II: Main Phase (N=186) | Wave II: Roll-In (N=30)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Wave I (N=40) | Wave II: Main Phase (N=186) | Wave II: Roll-In (N=30)
Atrial flutter (Cardiac disorders) | 4 (5) | 10 (10) | 0 (0)
Palpitation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erosive oesophagatis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oesophageal mucosa erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Mayocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 16 (16) | 6 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 5 (6) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 9 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 6 (7) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Apocrine breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0/4 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone loss (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Invertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Marrow hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Genital swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship will be determined prior to development of any manuscript. All information concerning the study, investigational medical device, sponsor operations, patent application, manufacturing processes, and basic scientific data supplied by the sponsor to the investigator and not previously published, are considered confidential and remain the sole property of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT04524364/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT04524364/SAP_001.pdf